CLINICAL TRIAL: NCT00553631
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) Enzyme Replacement Therapy Compared With Imiglucerase in Patients With Type I Gaucher Disease
Brief Title: Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) ERT Compared With Imiglucerase in Type I Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGT-GCB-039; 2007-002840-21 (EudraCT Number)
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease, Type 1
Keywords: Enzyme Replacement Therapy; Gaucher disease; glucocerebrosidase; beta-glucocerebrosidase; Acid beta-glucocerebrosidase; glucosylceramidase; D-glucosyl-N-acylsphingosine glucohydrolase; gene activation; human
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase; imiglucerase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GA-GCB (Experimental): VPRIV™ ,velaglucerase alfa
  Interventions: Biological: velaglucerase alfa
- imiglucerase (Active Comparator)
  Interventions: Biological: imiglucerase

INTERVENTIONS:
Biological: velaglucerase alfa — IV infusion, 60 U/kg every other week for 9 months
  Other Names: VPRIV™; gene-activated human glucocerebrosidase
  Arms: GA-GCB
Biological: imiglucerase — IV infusion, 60 U/kg every other week for 9 months
  Other Names: Cerezyme®
  Arms: imiglucerase

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to the deficiency of functional GCB, glucocerebroside accumulates within macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. The purpose of this non-inferiority study is to evaluate the efficacy and safety of GA-GCB (velaglucerase alfa) administered every other week in comparison to imiglucerase in treatment naive patients with type 1 Gaucher disease.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form, accounts for more than 90% of all cases and does not involve the CNS. Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Gene-Activated® human glucocerebrosidase (GA-GCB; velaglucerase alfa) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. GA-GCB (velaglucerase alfa) contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This study was designed to determine the efficacy and safety of GA-GCB (velaglucerase alfa) in comparison to imiglucerase in men, women, and children with Type 1 Gaucher disease.

ELIGIBILITY:
Inclusion Criteria

Includes:

* The patient has a documented diagnosis and clinical manifestation of type 1 Gaucher disease
* The patient is at least 2 years of age.
* The patient has not received treatment for Gaucher disease (investigational products, miglustat, or imiglucerase) within 12 months prior to study entry, as documented in the patient's medical history.
* Female patients of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study and must have negative results to a pregnancy test performed at the time of enrollment and as required throughout their participation in the study. Male patients must use a medically acceptable method of birth control throughout their participation in the study and must report their partner's pregnancy.
* The patient, the patient's parent(s) or legal guardian(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
* The patient must be sufficiently cooperative to participate in this clinical study as judged by the Investigator.

Exclusion Criteria

Includes:

* The patient has type 2 or 3 Gaucher disease or is suspected of having type 3 Gaucher disease.
* The patient has received treatment with any non-Gaucher disease-related investigational drug or device within the 30 days prior to study entry; such use during the study is not permitted.
* The patient is known to be positive for human immunodeficiency virus (HIV).
* The patient is known to be positive for hepatitis B and/or C.
* The patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
* The patient has a significant comorbidity(ies) that might affect study data or confound the study results (e.g., malignancies, primary biliary cirrhosis, autoimmune liver disease, etc.).
* The patient is unable to comply with the protocol, e.g., has a clinically relevant medical condition making implementation of the protocol difficult, has an uncooperative attitude, is unable to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the Investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01-29 (Actual); Primary Completion 2009-05-05 (Actual); Study Completion 2009-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Duke Children's Hospital & Health Center, Durham, North Carolina, United States
- Your Health S.A., Buenos Aires, Argentina
- India (3):
  - Malabar Institute of Medical Sciences Ltd., Calicut, Kerala
  - All India Institute of Medical Sciences, New Delhi
  - KEM Hospital Research Centre, Pune
- Shaare Zedek Medical Center, Jerusalem, Israel
- Sociedad Espanola de Socorros Mutuos, Asunción, Paraguay
- National Research Center for Haematology, Moscow, Russia
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- La Rabta Hospital, Tunis, Tunisia
- The Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Zimran A, Elstein D, Gonzalez DE, Lukina EA, Qin Y, Dinh Q, Turkia HB. Treatment-naive Gaucher disease patients achieve therapeutic goals and normalization with velaglucerase alfa by 4years in phase 3 trials. Blood Cells Mol Dis. 2018 Feb;68:153-159. doi: 10.1016/j.bcmd.2016.10.007. Epub 2016 Oct 21. PMID 27839979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in multiple sites from 29 January 2008 (first participant first enrolled) to 05 May 2009 (last participant completed).
Pre-assignment Details: Participants at least 2 years of age with type 1 Gaucher disease.Gaucher-disease-related anemia and at least 1 of the following: moderate splenomegaly, Gaucher-disease-related thrombocytopenia, readily palpable enlarged liver. Participants had not received treatment for Gaucher disease within 12 months prior to study entry.
Groups:
- Gene-Activated Human Glucocerebrosidase (GA-GCB): Velaglucerase alfa 60 unit per kilogram (U/kg) administered intravenously (IV) every other week for 39 weeks.
- Imiglucerase: Imiglucerase 60 U/kg administered IV every other week for 39 weeks.
Period: Overall Study
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Started | 17 (Intent-to-treat (ITT) population) | 17 (Intent-to-treat (ITT) population)
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gene-Activated Human Glucocerebrosidase (GA-GCB): Velaglucerase alfa 60 U/kg administered IV every other week for 39 weeks.
- Total: Total of all reporting groups
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants] — Age at time of consent
  Participants
    <=18 years | 4 | 5 | 9
    Between 18 and 65 years | 13 | 11 | 24
    >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 36 [7 to 60] | 27 [3 to 73] | 30.5 [3 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 8 | 8 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 1
  Paraguay | 3 | 2 | 5
  Argentina | 2 | 1 | 3
  Spain | 1 | 2 | 3
  Israel | 1 | 2 | 3
  Russian Federation | 2 | 2 | 4
  Tunisia | 4 | 2 | 6
  United Kingdom | 0 | 1 | 1
  India | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Month 9 in Hemoglobin (Hgb) Concentration for Each Treatment Group.
Time Frame: Baseline to Month 9
Population: Intent-to-treat (ITT) population comprised of all randomized participants who received at least 1 full or partial dose of study drug.
Measure: Mean (Standard Error); unit: gram per deciliter (g/dl)
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
gram per deciliter (g/dl) | 1.624 (0.223) | 1.488 (0.281)

2. Secondary Outcome: Change From Baseline to Month 9 in Platelet Counts for Each Treatment Group.
Description: Values shown are observed change from Baseline to Month 9.
Time Frame: Baseline to Month 9
Population: ITT population.
Measure: Mean (Standard Error); unit: 10^9 per liter (10^9/L)
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
10^9 per liter (10^9/L) | 110.41 (17.159) | 144.38 (22.76)

3. Secondary Outcome: Change From Baseline to Month 9 in Normalized Liver Volume (Percent (%) Body Weight) for Each Treatment Group.
Description: Values shown are observed change from Baseline to Month 9. Measured by Magnetic resonance imaging (MRI). Liver volume has been normalized for percent (%) body weight for each treatment arm. Liver size relative to body weight = (Liver volume [cubic centimeter (cc)]/Body weight [kg]*1000.
Time Frame: Baseline to Month 9
Population: ITT population.
Measure: Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
cubic centimeter (cm^3) | -1.31 (0.347) | -1.10 (0.182)

4. Secondary Outcome: Change From Baseline to Month 9 in Normalized Spleen Volume (Percent (%) Body Weight) for Each Treatment Group.
Description: Values shown are observed change from Baseline to month 9. Measured by Magnetic resonance imaging (MRI). Spleen volume was normalized for percent (%) of body weight for each treatment arm. Spleen size relative to body weight=(Spleen volume [cc]/Body weight [kg])*100.
Time Frame: Baseline to Month 9
Population: ITT population. Number of participants analyzed signifies participants evaluable for this outcome. Ten participants in each treatment group underwent splenectomy, and therefore, were excluded from the analysis.
Measure: Mean (Standard Error); unit: cm^3
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 7 | 7
cm^3 | -1.34 (0.424) | -2.46 (0.966)

5. Secondary Outcome: Change From Baseline to Month 9 in Plasma Chitotriosidase for Each Treatment Group.
Description: Values shown are observed change from Baseline to Month 9. Units of measure is defined as nanomole per milliliter per hour.
Time Frame: Baseline to Month 9.
Population: ITT population. Number of participants analyzed signifies participants evaluable for this outcome. Chitotriosidase levels were measured in 10 participants in the velaglucerase alfa group and 11 participants in the imiglucerase group.
Measure: Mean (Standard Error); unit: nanomole/milliliter/hour (nmol/mL/h)
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 10 | 11
nanomole/milliliter/hour (nmol/mL/h) | -34711.9 (6887.77) | -35109.5 (7310.22)

6. Secondary Outcome: Change From Baseline to Month 9 in Plasma Chemokine (C-C Motif) Ligand 18 (CCL18) for Each Treatment Group.
Description: Values shown are observed change from Baseline to Month 9.
Time Frame: Baseline to Month 9
Population: ITT population.
Measure: Mean (Standard Error); unit: nanogram per milliliter (ng/mL)
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
nanogram per milliliter (ng/mL) | -926.2 (113.29) | -1153.4 (269.63)

7. Secondary Outcome: Number of Participants Who Developed Antibody for Each Treatment Group.
Description: Measure type is actual number of participants who developed antibodies to treatment; GA-GCB or imiglucerase. Antibody detection was based upon serum samples collected at various time points throughout the study. Serum samples were screened using an enzyme-linked immunosorbent assay (ELISA) and positive antibody confirmation was determined using a radioimmunoprecipitation assay (RIP); positive samples were also tested for enzyme neutralizing activity. Participant samples were compared to internal assay controls (positive/negative), positive samples were determined based upon individual assay criteria.
Time Frame: Baseline to Month 9
Population: Safety population comprised of all randomized participants who received at least 1 full or partial dose of study drug.
Measure: Number; unit: participants
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
participants | 0 | 4

8. Secondary Outcome: Time to Response- Comparison of GA-GCB and Imiglucerase on the Earliest Time to Respond as Assessed Via Hemoglobin Concentration
Description: Time to response was defined as a ≥ 1 g/dL improvement in hemoglobin levels relative to Baseline. Units (%) correlates to the percentage of participants who had a change of ≥ 1 g/dL improvement in hemoglobin levels relative to Baseline during their participation in the study.
Time Frame: Response rate at Month 9 compared to Baseline
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Number analyzed (Participants) | 17 | 17
Percentage of participants | 92.9 | 100

ADVERSE EVENTS:
Time Frame: Adverse events (AE) monitored from time informed consent/assent obtained through 30 days after the last infusion. For participants who completed this study and elected to enroll in the long-term extension study, AEs were monitored through the Week 41.
Description: AE may have been discovered via observation, examination, questioning or complaint by participants.Unexpected laboratory values that became significantly out of range and determined to be clinically significant by the investigator could have been reported as AEs.Other AE were determined to be possibly/probably related to GA-GCB by the investigator.
Arm/Group | Gene-Activated Human Glucocerebrosidase (GA-GCB) | Imiglucerase
Serious Adverse Events (participants affected / at risk) | 3/17 | 0/17
Other Adverse Events (participants affected / at risk) | 16/17 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gene-Activated Human Glucocerebrosidase (GA-GCB) (N=17) | Imiglucerase (N=17)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Probably related
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) — Not related
Convulsions (Nervous system disorders) | 1 (1) | 0 (0) — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gene-Activated Human Glucocerebrosidase (GA-GCB) (N=17) | Imiglucerase (N=17)
Thrombocythaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (7) | 3 (6)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (11) | 3 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 2 (3)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (2)
Face oedema (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (3)
Feeling hot (General disorders) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (2)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Inflammatory pain (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Post-Traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis acute (Infections and infestations) | 1 (2) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0)
Infection parasitic (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (4) | 4 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants aged 2-4 years: 4 participants (23.5%) in imiglucerase group and 0 participants in GA-GCB group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.